CLINICAL TRIAL: NCT05076396
Title: Phase I, Open-label, Dose-escalating, Clinical and Pharmacokinetic Study of PM14 Administered Intravenously to Patients with Advanced Solid Tumors
Brief Title: PM14 Administered Intravenously to Patients with Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM14-A-001-17; 2017-001118-27 (EudraCT Number)
Record Dates: First submitted 2021-07-02; First posted 2021-10-13 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumor; PharmaMar; Cancer; PM14
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: First-in-human, open-label, dose-finding, phase I trial, using a classical 3+3 design followed by a continual reassessment method (CRM)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PM14 (Experimental): Patients will receive PM14 as an i.v. infusion in a total volume of 100 mL of 0.9% sodium chloride at the first three dose escalation levels. Thereafter, the volume of infusion can be increased to 250 mL.
  Interventions: Drug: PM14

INTERVENTIONS:
Drug: PM14 — PM14 drug product is provided as a sterile lyophilized powder for concentrate for solution for infusion with a strength of 5.0 mg of the active moiety. Patients will receive PM14 as an i.v. infusion in a total volume of 100 mL of 0.9% sodium chloride at the first three dose escalation levels. Thereafter, the volume of infusion can be increased to 250 mL.

SUMMARY:
Despite recent advances in the treatment of solid tumors in general, advanced (metastatic) disease remains mostly incurable and there is an urgent need to develop new therapeutic options for these patients, particularly investigational drugs with novel mechanisms of action. The investigation of new combination regimens of non-crossresistant agents with acceptable-and not completely overlapping-toxicities has been a major way to improve response rate and outcome of patients with advanced solid tumors.

DETAILED DESCRIPTION:
First-in-human, open-label, dose-finding, phase I trial, using a classical 3+3 design followed by a continual reassessment method (CRM).

Patients will be included in cohorts of a minimum of three or six patients to receive PM14 at successively increasing dose levels, starting at 0.25 mg/m^2 for the Days 1 and 8 schedule. For the Day 1 schedule, the starting dose will be 4.5 mg/m^2. Dose escalation will proceed only after all the patients fully evaluable for DLT included at one dose level have completed the first cycle (i.e., three weeks). Once the RD has been determined, expansion cohorts will be included to have a minimum of 20 fully evaluable patients per indication (tumor type) treated in the Expansion phase (regardless of the schedule administered), and thus have an adequate number of patients to assess safety. The indications of these patients will be chosen depending on the efficacy data obtained during dose escalation. Patients treated at the expansion cohorts will be evaluable by the Response Evaluation Criteria in Solid Tumors (RECIST v.1.1) and/or by serum markers only in patients with prostate cancer (prostate specific-antigen [PSA]) or ovarian cancer (carbohydrate antigen-125 [CA-125]) according to the Prostate-Specific Antigen Working Group Recommendations (PSAWGR) and the Gynecologic Cancer Intergroup (GCIG) specific criteria, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed and dated written informed consent (IC), obtained prior to any specific study procedure.
2. Age ≥18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤1
4. For the Dose escalation phase:

   Patients with pathologically confirmed diagnosis of advanced solid tumors for whom no curative standard therapy exists.

   For the Expansion phase:

   Patients with pathologically confirmed diagnosis of one of the following malignancies, for whom the standard of care therapies have failed, or are intolerant to standard of care therapies that are known to provide clinical benefit:
   1. Gastrointestinal tumors: colorectal cancer, gastric cancer.
   2. Sarcomas: liposarcoma, leiomyosarcoma, synovial sarcoma, Ewing's sarcoma.
   3. Tumors with deleterious germline BRCA mutation: epithelial ovarian cancer (including primary peritoneal and fallopian tube cancer), breast cancer, pancreatic cancer, prostate cancer, or any other malignancies.
   4. Epithelial ovarian cancer (including primary peritoneal and fallopian tube cancer) with no deleterious germline BRCA mutations or with unknown BRCA status.
   5. Adrenocortical carcinoma.
5. Patients included in the Expansion phase need to meet the following requirements regarding the maximum number of prior chemotherapy regimens (no limit for biological therapies):

   1. Gastrointestinal tumors: no more than three prior chemotherapy lines for colorectal cancer; and no more than two prior chemotherapy lines for gastric cancer.
   2. Sarcomas: no more than two prior chemotherapy lines for liposarcoma, leiomyosarcoma and synovial sarcoma; and no more than three prior chemotherapy lines for Ewing's sarcoma.
   3. Tumors with deleterious germline BRCA mutation: no more than three prior chemotherapy lines for breast cancer; and no more than two prior chemotherapy lines for prostate cancer, ovarian cancer, pancreatic cancer, gastric carcinoma, or any other malignancies.
   4. Epithelial ovarian cancer with unknown BRCA status or no deleterious germline BRCA mutations: no more than three prior chemotherapy lines.
   5. Adrenocortical cancer: no more than one prior chemotherapy line (excluding mitotane as single agent or associated with no chemotherapeutic agents).

   Note: for the purpose of this criterion, the following situations will be considered as one chemotherapy line:
   * Adjuvant chemotherapy; neoadjuvant chemotherapy; both adjuvant and neoadjuvant chemotherapy (except if time to relapse was >12 months, in which case it will not be considered as one line); and
   * Change of chemotherapy due to reasons other than PD, such as toxicity (in this case, the two lines will count as a single line).
6. Life expectancy ≥3 months.
7. Patients with measurable or non-measurable disease according to the RECIST v.1.1 are eligible during the dose escalation phase.
8. Patients included in the Expansion phase must have:

   1. Measurable disease according to the RECIST v.1.1 and/or evaluable disease by serum markers in case of prostate and ovarian cancer (according to the PSAWGR and the GCIG specific criteria, respectively).
   2. Confirmed progressive disease after last therapy at study entry.
9. Recovery to grade ≤1 from drug-related AEs of previous treatments, excluding alopecia and grade 1/2 asthenia or fatigue, according to the NCI-CTCAE v.4.
10. Laboratory values within seven days prior to first infusion:

    1. ANC ≥1.5 x 10^9/L, platelet count ≥100 x 10^9/L and hemoglobin ≥9 g/dL (patients may be transfused for anemia as clinically indicated prior to study entry).
    2. AST and ALT ≤3.0 x ULN.
    3. Total bilirubin ≤ULN (up to 1.5 x ULN for patients with Gilbert's syndrome).
    4. Creatinine clearance ≥30 mL/min (calculated using the Cockcroft and Gault's formula).
    5. Serum albumin ≥3 g/dL.
11. Wash-out periods:

    1. At least three weeks since the last chemotherapy (six weeks if therapy included nitrosoureas or systemic mitomycin C).
    2. At least four weeks since the last monoclonal antibody (MAb)-containing therapy or curative radiotherapy (RT).
    3. At least two weeks since the last biological/investigational single-agent therapy (excluding MAbs) and/or palliative RT (≤10 fractions or ≤30 Gy total dose).
    4. In patients with hormone-sensitive breast cancer progressing while on hormone therapy (except for luteinizing hormone-releasing hormone (LHRH) analogues in pre-menopausal women or megestrol acetate), all other hormonal therapies must be stopped at least one week before study treatment start.
    5. Castrate-resistant prostate cancer (CRPC) patients may continue receiving hormone therapy prior to and during study treatment.

Exclusion Criteria:

1. Concomitant diseases/conditions:

   1. Increased cardiac risk:

      * Uncontrolled arterial hypertension despite optimal management (≥160/100 mmHg).
      * Presence of clinically relevant valvular disease.
      * History of long QT syndrome.
      * Corrected QT interval (QTcF, Fridericia correction) ≥450 msec on screening electrocardiogram (ECG).
      * History of ischemic heart disease, including myocardial infarction, angina, coronary arteriography or cardiac stress testing with findings consistent with coronary occlusion or infarction ≤6 months prior to study entry.
      * History of heart failure or left ventricular dysfunction (left ventricular ejection fraction [LVEF] below normal values) by multiple-gated acquisition scan (MUGA) or echocardiography (ECHO).
      * ECG abnormalities, including any of the following: left bundle branch block, right bundle branch block with left anterior hemiblock, second (Mobitz II) or third degree atrioventricular block.
      * Symptomatic arrhythmia (excluding anemia-related sinusal tachycardia grade ≤2) or any arrhythmia requiring ongoing treatment, and/or prolonged QT-QTc grade ≥2; or presence of unstable atrial fibrillation. Patients with stable atrial fibrillation on treatment are allowed provided they do not meet any other cardiac or prohibited drug exclusion criterion.
      * Clinically significant resting bradycardia (<50 beats per minute).
      * Concomitant medication with risk of inducing torsades de pointes, which cannot be discontinued or switched to an alternative drug prior to start PM14 dosing.
      * Use of a cardiac pacemaker.
   2. Active infection requiring systemic treatment.
   3. Known human immunodeficiency virus (HIV) or known hepatitis C virus (HCV) infection or active hepatitis B.
   4. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study (e.g., COVID-19).
2. Symptomatic, high dose steroid-requiring, and progressing central nervous system (CNS) disease. Exceptions will be made for (i) patients who have completed radiotherapy at least four weeks prior to inclusion (asymptomatic, non-progressing patients taking steroids in the process of already being tapered within two weeks prior to inclusion), and (ii) patients with asymptomatic brain metastasis without need for radiotherapy or steroids.
3. Patients with carcinomatous meningitis regardless of clinical stability.
4. Prior bone marrow or stem cell transplantation, or radiation therapy in more than 35% of bone marrow.
5. Prior treatment with trabectedin or Lurbinectedin (PM01183) within six months prior to onset of study treatment.
6. Use of (strong or moderate) inhibitors or strong inducers of CYP3A4 activity within two weeks prior to the first infusion of PM14.
7. Known hypersensitivity to any of the components of the drug product
8. Limitation of the patient's ability to comply with the treatment or to follow the protocol procedures.
9. Pregnant or lactating women. Women of childbearing potential (WOCBP) must agree to use an effective contraception method to avoid pregnancy during trial treatment and for at least six months after the last infusion. Fertile male patients must agree to refrain from fathering a child or donating sperm and to use an effective contraception method during treatment and for four months after the last infusion. WOCBP who are partners of fertile male patients must use an effective contraception method during the patients' treatment and for four months after the last infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-09-06 (Actual); Primary Completion 2025-08-13 (Estimated); Study Completion 2025-08-13 (Estimated)

PRIMARY OUTCOMES:
Patients with dose limiting toxicities | At cycle 2 (21-days cycle)
  To identify the dose limiting toxicities (DLTs), and to determine the maximun tolerated dose (MTD) and the recommended dose (RD) of PM14 administered i.v. on two days (Day 1 and Day 8) or on Day 1 only, both every three weeks (q3wk) over three hours to patients with advanced solid tumors.
Overall response rate | At cycle 2 (21-days cycle)
  To confirm the recommended dose (RD) determined during the Dose escalation phase, and to evaluate the antitumor activity of PM14 in terms of overall response rate (ORR), according to the Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1, and/or serum markers as appropriate, in patients with selected advanced solid tumors.
Overall response rate | At cycle 4 (21-days cycle)
  To confirm the recommended dose (RD) determined during the Dose escalation phase, and to evaluate the antitumor activity of PM14 in terms of overall response rate (ORR), according to the Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1, and/or serum markers as appropriate, in patients with selected advanced solid tumors.
Overall response rate | At cycle 6 (21-days cycle)
  To confirm the recommended dose (RD) determined during the Dose escalation phase, and to evaluate the antitumor activity of PM14 in terms of overall response rate (ORR), according to the Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1, and/or serum markers as appropriate, in patients with selected advanced solid tumors.
Overall response rate | Through study completion up to Cycle 9
  To confirm the recommended dose (RD) determined during the Dose escalation phase, and to evaluate the antitumor activity of PM14 in terms of overall response rate (ORR), according to the Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1, and/or serum markers as appropriate, in patients with selected advanced solid tumors.

SECONDARY OUTCOMES:
Clinical Benefit Rate | Through study completion up to Cycle 9
  Clinical benefit rate in each tumor type is defined as the percentage of patients with a confirmed response (either complete response or partial response) according to the RECIST v.1.1 and/or by serum markers or with stable disease (SD) ≥4 months
Progression-free Survival | From the date of first infusion of study treatment to the date of first documented progression or date of death from any cause, assessed up to 72 months
  Progression-free survival (PFS) is defined as the time from the date of first infusion of study treatment to the date of documented progression or death (due to any cause). If progression or death has not occurred at the time of the analysis, the PFS will be censored on the date of last tumor evaluation.
Duration of Response | From the date of the first documentation of response to the date of first PD or further therapy or death, assessed up to 72 months
  Duration of response (DoR) is defined as the time between the date of first documentation of response to the date of documented progression or death.
Incidence of Treatment-Emergent Adverse Events | From the date of first infusion of study treatment to the date of study termination, assessed up to 72 months
  Patients will be evaluable for safety if they have received at least one partial infusion of PM14. Adverse events (AEs) will be graded according to the NCI-CTCAE v.4. Additionally, treatment related discontinuations and treatment compliance (dose reduction, skipped doses and/or treatment delays due to AEs) will be described.
Pharmacokinetic: Maximum Plasma Concentration (Cmax) | At the end of Cycle 1 (each cycle is 21 days)
  Pharmacokinetic analyses will be evaluated in plasma and urine by standard noncompartmental analysis. Compartmental modeling may be performed if appropriate.
Pharmacokinetic: Area Under The Concentration-time Curve (AUC) | At the end of Cycle 1 (each cycle is 21 days)
  Pharmacokinetic analyses will be evaluated in plasma and urine by standard noncompartmental analysis. Compartmental modeling may be performed if appropriate.
Pharmacogenetic | At the end of Cycle 1 (each cycle is 21 days)
  To evaluate Pharmacogenetic (PGt) in germline DNA by the presence or absence of PGt polymorphisms in genes relevant for PM14 disposition
Pharmacogenomic: Number of patients with RNA/protein expression | At the end of Cycle 1 (each cycle is 21 days)
  To conduct an exploratory Pharmacogenomic analysis in tumor tissue samples and ctDNA of patients treated with PM14. Quantitation of mRNA expression of selected genes involved in DNA repair mechanisms or related to the mechanism of action of PM14 by qRT-PCR. Quantitation of protein expression of these genes by IHC, in tumor tissue samples.
Pharmacogenomic: Number of patients with Polymorphisms | At the end of Cycle 1 (each cycle is 21 days)
  To conduct an exploratory Pharmacogenomic analysis in tumor tissue samples and ctDNA of patients treated with PM14.
  Evaluate the presence or absence of polymorphisms in genes relevant for PM14 disposition
Pharmacogenomic: Number of patients with Mutations | At the end of Cycle 1 (each cycle is 21 days)
  To conduct an exploratory Pharmacogenomic analysis in tumor tissue samples and ctDNA of patients treated with PM14. The mutational status of genes wil also be analyzed

CONTACTS AND LOCATIONS:
Locations (9):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas
- Gustave Roussy, Villejuif, París, France
- Spain (6):
  - Hospital Universitari Vall d'Hebron, Barcelona, Catalonia
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Clinica Universidad de Navarra, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid, Madrid